CLINICAL TRIAL: NCT02429232
Title: A One-year Randomized Controlled Trial Evaluating the Impact of Pioglitazone Versus Linagliptin on Bone Turnover Markers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201312136MIND
Record Dates: First submitted 2015-04-07; First posted 2015-04-29 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis; Diabetes Mellitus
Keywords: Pioglitazone; Linagliptin; Diabetes mellitus; Diabetic macular edema; Kidney
MeSH Terms: conditions — Osteoporosis; Diabetes Mellitus | interventions — Pioglitazone; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Experimental): Pioglitazone 30 mg once daily will be administered orally for total 48 weeks.
  Interventions: Drug: Pioglitazone
- Linagliptin (Active Comparator): Linagliptin 5 mg once daily will be administered orally for total 48 weeks.
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30mg/tablet once daily
  Other Names: Actos
  Arms: Pioglitazone
Drug: Linagliptin — Linagliptin 5mg/tablet once daily
  Other Names: Trajenta
  Arms: Linagliptin

SUMMARY:
Diabetes mellitus is a common disease with much impact on human's health and is related to osteoporosis. But the mechanism remains unclear. The foreign researches revealed thiazolidinedione (TZD) would increase the risk of osteoporosis and bone fracture, specially elderly women. However, it is still controversial in terms of the youth and men. In Taiwan,there is few related study to analyze the relationship between TZD and steoporosis.

This is a multicenter randomized controlled study.

DETAILED DESCRIPTION:
Diabetes mellitus is a common disease with much impact on human's health and is related to osteoporosis. But the mechanism remains unclear. The foreign researches revealed thiazolidinedione (TZD) would increase the risk of osteoporosis and bone fracture, especially elderly women. However, it is still controversial in terms of the youth and men. In Taiwan, there is few related study to analyze the relationship between TZD and osteoporosis.

This is a multicenter randomized controlled study.This study will recruit adult (age ³40 years) type 2 diabetes patients who is on metformin (³1500mg/day) currently with recent HbA1c between 7.0~8.5%.Patient who has history of macular edema, congestive heart failure (NYHA Fc III, IV), chronic renal failure (stage IV, V), AST or ALT above 2.5 times upper limit, Medical history of endocrinopathies, osteoporosis with bone fracture, cancer will be excluded. Current bone fracture undergoing treatment, pregnancy, breast feeder will also be excluded.

This is a 3-year project and will enroll 160 eligible volunteers who are to randomized into group A and B (80 in each). During the next 48 weeks group A and B will receive metformin+pioglitazone and metformin+linagliptin respectively. Blood sugar, renal, and liver functions will be examined every 12 weeks. Calcium, phosphorus, vitamin D level, and bone turnover markers (N-terminal propeptide of type 1 procollagen, bone-specific alkaline phosphatase, osteocalcin, serum C- telopeptide, type 5 tartrate resistant acid phosphatase (TRAP), pyridinoline and deoxypyridinoline crosslinks) will be checked each 6 months.

All the blood samples will be sent to one core laboratory center. The within-group differences will be examined by repeated-measure ANOVA. The between-group differences will be examined by Student's t test.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or females ≥ 40 years of age at Visit 1and females in postmenopause for one year
* Documentation of type 2 diabetes mellitus as evidenced by one or more of the following criteria:

  1. With typical symptoms and random blood sugar ≥ 200 mg/dl
  2. 8-hour fasting blood sugar ≥ 126 mg/dl
  3. Oral glucose tolerance test ≥ 200 mg/dl
  4. HbA1c≥ 6.5%
* Only receiving oral anti-diabetic drugs (excluding TZDs or DPP-4 inhibitors) till visit 1 at least 3 months, and the HbA1c is between 7.0~8.5 % in recent 3 months.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* DM on oral anti-diabetic drugs less than 3 months.
* Receiving treatment of TZDs or DPP-4 inhibitors prior to this study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* AST, ALT over 2.5 times of the upper limit.
* Chronic kidney disease, stage 4 and 5.
* Congestive heart failure, NYHA class III, IV
* History of osteoporosis.
* History of diseases known to affect bone metabolism:

Abnormal thyroid function or history of hyperthyroidism, Cushing's syndrome, hypogonadism, acromegaly, history of hypopituitarism or status post pituitary surgery and/or radiotherapy, hematopoietic disorders.

* History of moderate to severe Diabetic macular edema (DME)
* History of moderate to severe diabetic retinopathy.
* History of fracture over lumbar spine or hip joint or femoral head or forearm or any site of bone fracture undergoes treatment currently.
* Who had taken any of the following medications prior to screening:

Corticosteroid, heparin, anticonvulsants, aluminum-containing antacid, proton pump inhibitor, immunosuppressant user within 3 months. Bisphosphonate, systemic fluoride treatment, PHT analogue, calcitonin, Denosumab, Strontium ranelate, hormone replacement therapy (androgen/estrogen/progesterone, thyroxine, growth hormone), selective estrogen receptor modulator /SERM (Tamoxifene, Raloxifene), selective tissue estrogenic activity regulator /STEAR (Tibolone), aromatase inhibitors within 1 year.

* History of cancer.
* Bed-ridden patients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in bone turnover markers | Screen, Week 24, 48
  The primary objective is to assess the effect of TZD on skeleton as measured bone turnover markers over the 12 months treatment period.

SECONDARY OUTCOMES:
Change from baseline in Estimated glomerular filtration rate( eGFR) | Screen, Week 24, 48
  The objective is to assess the effect of TZD on kidney by measurement of Estimated glomerular filtration rate( eGFR) over the 12 months treatment period.
Change from baseline in renal function-serum Creatinine (Cr) level | Screen, Week 24, 48
  The secondary objective is to assess the effect of TZD on kidney by measurement of doubling time of serum Creatinine (Cr) level and urine biomarkers over the 12 months treatment period.
Change from baseline in renal function-Urine Albumin-to-Creatinine Ratio(UACR) | Screen, Week 24, 48
  The secondary objective is to assess the effect of TZD on kidney by measurement of doubling time of Urine Albumin-to-Creatinine Ratio(UACR) and urine biomarkers over the 12 months treatment period.
Change from baseline in urine biomarkers | Screen, Week 24, 48
  The secondary objective is to assess the effect of TZD on kidney by measurement of urine biomarkers over the 12 months treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hsiao Tseng, MD, PhD, Principal Investigator — Department of Medicine,National Taiwan University Hospital